CLINICAL TRIAL: NCT00082498
Title: Phase II, Randomized, Double-Blind Study of the Safety and Efficacy of Vicriviroc (An Orally Administered HIV-1 Entry Inhibitor) in HIV-Infected, Treatment-Experienced Subjects
Brief Title: Safety and Effectiveness of the Oral HIV Entry Inhibitor Vicriviroc in HIV Infected Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A5211; 10097 (Registry Identifier: DAIDS ES); ACTG A5211; 5K24AI051966-03 (NIH)
Record Dates: First submitted 2004-05-11; First posted 2004-05-12 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: SCH-D; Schering D; Treatment Experienced; Entry Inhibitors; Fusion Inhibitors; Vicriviroc
MeSH Terms: conditions — HIV Infections | interventions — vicriviroc

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1 (Placebo Comparator): Group 1 will receive placebo
  Interventions: Drug: Placebo
- 2 (Experimental): Group 2 will receive 5 mg vicriviroc daily
  Interventions: Drug: SCH-D (vicriviroc)
- 3 (Experimental): Group 3 will receive 10 mg vicriviroc daily
  Interventions: Drug: SCH-D (vicriviroc)
- 4 (Experimental): Group 4 will receive 15 mg vicriviroc daily
  Interventions: Drug: SCH-D (vicriviroc)

INTERVENTIONS:
Drug: SCH-D (vicriviroc) — Group 2 will receive 5 mg vicriviroc daily; Group 3 will receive 10 mg vicriviroc daily; and Group 4 will receive 15 mg vicriviroc daily. If at or after Week 16 a participant's viral load has not met certain criteria, a dose increase of vicriviroc may occur and the participant will enter Step 2. As of 10/12/05, patients in Group 2 and any patients who entered Step 2 following virologic failure in Step 1 will be unblinded and offered either 15 mg vicriviroc daily through this study or the option of seeking alternative treatment.
  Arms: 2; 3; 4
Drug: Placebo — Patients in Group 1 will receive placebo.
  Arms: 1

SUMMARY:
New treatment options are critical for treatment-experienced HIV infected patients with drug resistance. HIV entry inhibitors have been shown effective in patients with resistance to other anti-HIV drugs. This study will test the safety and effectiveness of three different doses of vicriviroc (formerly known as Schering D, SCH-D, or SCH 417690) in HIV infected patients.

DETAILED DESCRIPTION:
Vicriviroc is an oral HIV-1 entry inhibitor that targets the CCR5 receptor of T cells. Vicriviroc has been shown safe, well-tolerated, and active in Phase I clinical trials in treatment-naive HIV infected patients. The goal of this study is to evaluate the antiretroviral activity of three dose levels of vicriviroc in HIV infected, treatment-experienced patients who are failing their current ritonavir-containing antiretroviral therapy (ART).

The study will last at least 48 weeks, but no more than 5 years. There are 3 steps in this study. Patients will be randomly assigned to one of 4 groups. Group 1 will receive placebo; Group 2 will receive 5 mg vicriviroc daily; Group 3 will receive 10 mg vicriviroc daily; and Group 4 will receive 15 mg vicriviroc daily. If at or after Week 16 a participant's viral load has not met certain criteria, a dose increase of vicriviroc may occur and the participant will enter Step 2. As of 10/12/05, patients in Group 2 and any patients who entered Step 2 following virologic failure in Step 1 will be unblinded and offered either 15 mg vicriviroc daily through this study or the option of seeking alternative treatment. All patients will continue their current ART (not provided by the study). After two weeks, patients will receive ART optimized by the results of genotypic/phenotypic testing performed at study screening. All participants who have received or are receiving vicriviroc will enter Step 3 and be followed for an additional 4 years. Participants who complete the study may be eligible to receive vicriviroc through a rollover study sponsored by Schering-Plough, the drug's manufacturer.

Physical exams and blood collection will occur at study entry, Day 4, and Weeks 1, 2, 4, 8, 12, 16, 20, 24, 32, 40, and 48. Additionally, blood will be drawn twice, at least 2 hours apart, at both Weeks 2 and 8 for vicriviroc pharmacokinetic analysis. Patients will undergo an electrocardiogram (EKG) at Weeks 2, 8, 24, and 48. Patients will be assessed for peripheral neuropathy at study entry and Weeks 24 and 48, and will be asked to complete an adherence questionnaire at entry and Weeks 2, 8, 16, 24, 32, 40, and 48. For Step 3 participants undergoing follow-up, physical exams and blood work will occur every 6 months for 4 years.

Five participants currently enrolled at four sites that are no longer receiving funding and who will not be transferred or redirected to a site within their proximity will be subject to the following changes. There will no longer be follow-up visits per the schedule of events described in the protocol. Instead, participants will have their follow-up limited to self-report through telephone interviews to ascertain vital status, occurrence of malignancies (if any), and collection of information such as HIV-1 RNA and CD4 cell count. For these participants only, the HIV-1 RNA and CD4 cell count will be done as part of the participant's clinical care and will not be paid for by the study. The follow-up telephone interviews will be conducted at six-month intervals using the script provided by the study team.

ELIGIBILITY:
Note: This study was closed to screening on 09/20/05 and to enrollment on 10/20/05.

Inclusion Criteria for Step 1:

* HIV infected
* Experiencing virologic failure on current ART regimen
* Current ART regimen contains ritonavir (100 to 800 mg/day) and has been stable for at least 8 weeks prior to study entry. If amprenavir or fosamprenavir is part of the regimen, 200 to 800 mg/day ritonavir must be used for at least 2 weeks prior to study entry.
* Experienced virologic failure on at least one ART regimen containing 3 or more drugs prior to current failing regimen
* CD4 count of 50 cells/mm3 or more within 6 weeks prior to study entry
* HIV viral load of 5,000 copies/ml or more within 6 weeks prior to study entry
* HIV strain of R5-only phenotype within 6 weeks prior to study entry
* Willing to use acceptable forms of contraception
* Able and willing to adhere to study dose and visit schedules

Inclusion Criteria for Step 2:

* HIV viral load not suppressed by at least 1log10 below baseline viral load by Week 16 or after
* QTc interval on EKG less than 500 msec, and less than 60 msec increase from baseline within 14 days of Step 2 entry

Inclusion Criteria for Step 3:

* Use of vicriviroc in Step 1 or 2 of this study or the Schering rollover study. Participants who are currently not taking vicriviroc are eligible.

Exclusion Criteria for Step 1:

* Hepatitis C antibody and RNA positive
* Hepatitis B surface antigen positive
* Efavirenz or nevirapine use within 8 weeks of study entry
* Vaccination within 2 weeks prior to study screening
* Investigational agents within 30 days prior to study entry
* Systemic cancer chemotherapy or other systemic cytotoxic agents within 30 days prior to study entry
* Immunosuppressants within 30 days prior to study entry. Systemic corticosteroids at replacement doses (10 mg/day prednisone or less) are not excluded.
* Immunomodulators within 30 days prior to study entry
* Considered at risk for seizure: history of seizure, recent history of head trauma with loss of consciousness, central nervous system (CNS) tumors, or other CNS problems that, in the opinion of the investigator, pose increased risk for seizure
* Medications to prevent seizures or with the potential to cause seizures within 30 days prior to study entry
* Allergy to SCH 417690 or its components
* Alcohol or drug abuse that, in the opinion of the investigator, would interfere with the study
* Serious illness requiring systemic treatment or hospitalization. A patient who is clinically stable on therapy is not excluded.
* Any clinically significant disease or condition that, in the opinion of the investigator, may interfere with the study
* Require certain medications
* Pregnancy or breastfeeding

Exclusion Criteria for Step 2:

* Have X4 or X4/R5 tropic virus, as determined by the HIV-1 coreceptor tropism assay
* Intend to use efavirenz or nevirapine in background ART regimen
* Allergy to vicriviroc or its formulations
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2004-05; Primary Completion 2005-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Change in HIV-1 viral load | From baseline to Day 14

SECONDARY OUTCOMES:
Safety and tolerability | Throughout the study
Virologic and immunologic outcomes | Throughout the study
Clinical outcomes | Throughout the study
Pharmacokinetic outcomes | At Weeks 2 and 8
Viral coreceptor phenotype | At study entry, Day 4, and Weeks 1, 2, 4, 8, 12, 16, 20, 24, 32, 40, and 48
Adherence measures | At study entry and Weeks 2, 8, 16, 24, 32, 40, and 48

CONTACTS AND LOCATIONS:
Overall Officials: Roy M. Gulick, MD, MPH, Study Chair — Cornell HIV Clinical Trials Unit; Charles Flexner, MD, Study Chair — Johns Hopkins University Hospital; Daniel Kuritzkes, MD, Study Chair — Harvard Medical School, Partners AIDS Research Center
Locations (30):
- United States (30):
  - UCLA CARE Center CRS, Los Angeles, California
  - Stanford AIDS Clinical Trials Unit CRS, Palo Alto, California
  - UCSD Antiviral Research Center CRS, San Diego, California
  - Ucsf Hiv/Aids Crs, San Francisco, California
  - Santa Clara Valley Med. Ctr., San Jose, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Georgetown University CRS (GU CRS), Washington D.C., District of Columbia
  - The Ponce de Leon Center CRS, Atlanta, Georgia
  - Rush University CRS, Chicago, Illinois
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Massachusetts General Hospital CRS (MGH CRS), Boston, Massachusetts
  - Brigham and Women's Hospital Therapeutics Clinical Research Site (BWH TCRS) CRS, Boston, Massachusetts
  - Bmc Actg Crs, Boston, Massachusetts
  - Washington University Therapeutics (WT) CRS, St Louis, Missouri
  - Beth Israel Med. Ctr., ACTU, New York, New York
  - Weill Cornell Chelsea CRS, New York, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Weill Cornell Uptown CRS, New York, New York
  - Trillium Health ACTG CRS, Rochester, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Chapel Hill CRS, Chapel Hill, North Carolina
  - Case CRS, Cleveland, Ohio
  - MetroHealth CRS, Cleveland, Ohio
  - Ohio State University CRS, Columbus, Ohio
  - Penn Therapeutics, CRS, Philadelphia, Pennsylvania
  - University of Pittsburgh CRS, Pittsburgh, Pennsylvania
  - The Miriam Hospital Clinical Research Site (TMH CRS) CRS, Providence, Rhode Island
  - Vanderbilt Therapeutics (VT) CRS, Nashville, Tennessee
  - Univ. of Texas Medical Branch, ACTU, Galveston, Texas
  - University of Washington AIDS CRS, Seattle, Washington

REFERENCES:
- [Background] Marks K, Gulick RM. New antiretroviral agents for the treatment of HIV infection. Curr HIV/AIDS Rep. 2004 Jun;1(2):82-8. doi: 10.1007/s11904-004-0012-0. PMID 16091227
- [Background] Meanwell NA, Kadow JF. Inhibitors of the entry of HIV into host cells. Curr Opin Drug Discov Devel. 2003 Jul;6(4):451-61. PMID 12951808
- [Background] Reeves JD, Piefer AJ. Emerging drug targets for antiretroviral therapy. Drugs. 2005;65(13):1747-66. doi: 10.2165/00003495-200565130-00002. PMID 16114975
- [Background] Schurmann D et al. SCH D: Antiviral activity of a CCR5 receptor antagonist. 11th Conf Retro and Opportun Infect. 2004 Feb 8-11 (abstract no 140LB).
- [Background] Shaheen F, Collman RG. Co-receptor antagonists as HIV-1 entry inhibitors. Curr Opin Infect Dis. 2004 Feb;17(1):7-16. doi: 10.1097/00001432-200402000-00003. PMID 15090884
- [Background] Strizki JM, Tremblay C, Xu S, Wojcik L, Wagner N, Gonsiorek W, Hipkin RW, Chou CC, Pugliese-Sivo C, Xiao Y, Tagat JR, Cox K, Priestley T, Sorota S, Huang W, Hirsch M, Reyes GR, Baroudy BM. Discovery and characterization of vicriviroc (SCH 417690), a CCR5 antagonist with potent activity against human immunodeficiency virus type 1. Antimicrob Agents Chemother. 2005 Dec;49(12):4911-9. doi: 10.1128/AAC.49.12.4911-4919.2005. PMID 16304152
- [Result] Wilkin TJ, Su Z, Kuritzkes DR, Hughes M, Flexner C, Gross R, Coakley E, Greaves W, Godfrey C, Skolnik PR, Timpone J, Rodriguez B, Gulick RM. HIV type 1 chemokine coreceptor use among antiretroviral-experienced patients screened for a clinical trial of a CCR5 inhibitor: AIDS Clinical Trial Group A5211. Clin Infect Dis. 2007 Feb 15;44(4):591-5. doi: 10.1086/511035. Epub 2007 Jan 17. PMID 17243065
- [Derived] Wilkin TJ, Su Z, Krambrink A, Long J, Greaves W, Gross R, Hughes MD, Flexner C, Skolnik PR, Coakley E, Godfrey C, Hirsch M, Kuritzkes DR, Gulick RM. Three-year safety and efficacy of vicriviroc, a CCR5 antagonist, in HIV-1-infected treatment-experienced patients. J Acquir Immune Defic Syndr. 2010 Aug;54(5):470-6. doi: 10.1097/qai.0b013e3181e2cba0. PMID 20672447
- [Derived] Tsibris AM, Paredes R, Chadburn A, Su Z, Henrich TJ, Krambrink A, Hughes MD, Aberg JA, Currier JS, Tashima K, Godfrey C, Greaves W, Flexner C, Skolnik PR, Wilkin TJ, Gulick RM, Kuritzkes DR. Lymphoma diagnosis and plasma Epstein-Barr virus load during vicriviroc therapy: results of the AIDS Clinical Trials Group A5211. Clin Infect Dis. 2009 Mar 1;48(5):642-9. doi: 10.1086/597007. PMID 19191652